CLINICAL TRIAL: NCT01228864
Title: Brody Belt - Alternative Method of Securing a Patient's Urinary Drainage Bag
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 153209
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Quality of Life
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brody Belt (Experimental)
  Interventions: Procedure: quality of life
- Conventional Urinary Drainage bag (Active Comparator)
  Interventions: Procedure: Quality of life

INTERVENTIONS:
Procedure: quality of life — survey
  Arms: Brody Belt
Procedure: Quality of life
  Arms: Conventional Urinary Drainage bag

SUMMARY:
The Brody belt may help improve quality of life in patients using urinary drainage bags. PURPOSE: This clinical trial studies the Brody belt in improving the quality of life in patients using urinary drainage bags.

ELIGIBILITY:
Inclusion Criteria:

->18 years old

-All patients in the urology clinic at Roswell Park who currently use a urinary drainage bag for a period of at least 7 days prior to signing consent for the study and who are expected to use a urinary drainage tube for an additional period of 4 weeks or more based on the diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09-22 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Khurshid Guru, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States